CLINICAL TRIAL: NCT01355835
Title: Combined STN/SNr-DBS for the Treatment of Refractory Gait Disorders in Parkinson's Disease: Design of a Two-armed Double-blind Cross-over Study
Brief Title: Combined STN/SNr-DBS for the Treatment of Refractory Gait Disorders in Parkinson's Disease
Acronym: STN/SNr
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Daniel Weiss, MD, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKF 259-0-0
Record Dates: First submitted 2011-05-13; First posted 2011-05-18 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; gait; deep brain stimulation; substantia nigra pars reticulata; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- [STNmono] (Active Comparator): Conventional stimulation on subthalamic contacts
  Interventions: Device: deep brain stimulation (ACTIVA PC, Medtronic)
- [STN+SNr] (Experimental): Combined subthalamic and nigral stimulation
  Interventions: Device: deep brain stimulation (ACTIVA PC, Medtronic)

INTERVENTIONS:
Device: deep brain stimulation (ACTIVA PC, Medtronic) — High frequent deep brain stimulation with variable (best individual) stimulation on subthalamic contacts and standard parameters on nigral contacts (125 Hz, 60µs, best individual amplitude)
  Other Names: Neurostimulation with ACTIVA PC, Medtronic

SUMMARY:
12 patients with idiopathic Parkinson's disease and refractory gait disturbances under best individual subthalamic nucleus stimulation and dopaminergic medication will be included into this randomised double-blind cross-over two-armed clinical trial. The treatment consists of two different stimulation settings using (i) conventional stimulation of the subthalamic nucleus [STNmono] and (ii) combined stimulation of distant electrode contacts located in the subthalamic nucleus and caudal border zone of STN and substantia nigra pars reticulata [STN+SNr].

DETAILED DESCRIPTION:
A composite 'axial score' including the major clinical and anamnestic items on gait, posture and balance function from UPDRSII (items 13-15) and UPDRS III (items 27-31) constitutes the primary outcome measure. Secondary outcome measures include specified clinical and anamnestic assessments on freezing of gait, balance, quality of life, non-motor symptoms, impulsivity, impulse control and neuropsychiatric symptoms. The aim of the present trial is to investigate the efficacy and safety of combined stimulation on subthalamic and nigral electrode contacts [STN+SNr] in refractory hypokinetic gait disturbances compared with [STNmono] (active comparator). The results will clarify, whether the combined [STN+SNr] stimulation improves otherwise refractory gait disturbances in PD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age: between 18 and 80 years
* Idiopathic Parkinson's disease (according to the "British Brain Bank criteria" (Hughes, 1992) including genetic forms and therapy with STN-DBS (ACTIVA pulse generators) at least six months from surgery
* Optimized subthalamic stimulation at study enrolment (refer 'treatment' section)
* Gait disturbance refractory on best individual STN-DBS (STNmono) and dopaminergic therapy: 'gait score' in the best clinical [MedOn/STNmono] condition ≥ 12
* Clinical and image-guided (and facultatively electrophysiological) confirmation of (i) one of the two rostral contacts of the quadripolar electrode localized in the STN area, and (ii) the caudal contacts in the border zone of STN and SNr.
* Dopaminergic medication constant for at least four weeks prior to study enrolment
* Disease duration ≥ 5 years

Exclusion Criteria:

* Cognitive impairment (Mini Mental State Exam < 25)
* Participation in other clinical trials within the past three months and during enrolment in our study
* Suicidality, Psychosis
* Other severe pathological chronic condition that might confound treatment effects or interpretation of the data
* Pregnancy
* Acute adverse events from stimulation on contacts in the caudal STN / SNr border interfering with the intended stimulation protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
'Axial score' | Three weeks after active treatment (STN vs. STN+SNr), respectively
  The composite 'axial score' is built by 8 items from the UPDRS II and III, all 5-point rated (0 to 4) representing increasing levels of pathology. The 'axial score' will be scored by the sum of the ratings across the 8 items (Range 0 to 32). As change in UPDRS scores is a common primary efficacy outcome measure in Parkinson's disease and only items of the original UPDRS are required for the definition of the primary endpoint, the statistical evaluation methods should be based on the psychometric validation of the UPDRS and no own validation studies are necessary.
  Safety: falls

SECONDARY OUTCOMES:
CAPSIT-PD | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Freezing of gait assessment course | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Freezing of gait questionnaire | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Berg Balance Scale | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Non-motor symptoms scale | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Non-motor symptoms quest | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Beck's depression scale index | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Minnesota Impulsive Disorders Interview | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
Barratt Impulsiveness Scale | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
UPDRS I-IV | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively
PDQ-39 | At baseline and three weeks after active treatment (STN vs. STN+SNr), respectively

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Principal Investigator — Center of Neurology and Hertie Institute for Clinical Brain Research, and Department for Neurodegenerative Diseases, University of Tübingen; Rejko Krüger, MD, Principal Investigator — Center of Neurology and Hertie Institute for Clinical Brain Research, and Department for Neurodegenerative Diseases, University of Tübingen
Locations (1):
- Center of Neurology and Hertie Institute for Clinical Brain Research, and Department for Neurodegenerative Diseases, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Weiss D, Breit S, Wachter T, Plewnia C, Gharabaghi A, Kruger R. Combined stimulation of the substantia nigra pars reticulata and the subthalamic nucleus is effective in hypokinetic gait disturbance in Parkinson's disease. J Neurol. 2011 Jun;258(6):1183-5. doi: 10.1007/s00415-011-5906-3. Epub 2011 Feb 2. No abstract available. PMID 21287187
- [Derived] Weiss D, Wachter T, Meisner C, Fritz M, Gharabaghi A, Plewnia C, Breit S, Kruger R. Combined STN/SNr-DBS for the treatment of refractory gait disturbances in Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2011 Oct 11;12:222. doi: 10.1186/1745-6215-12-222. PMID 21989388